CLINICAL TRIAL: NCT00340379
Title: A Comparison of Two Different Treatments for Major Depression With Psychotic Features: Ziprasidone vs. Combined Sertraline and Haloperidol
Brief Title: Ziprasidone vs. Sertraline/Haloperidol in Psychotic Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry); National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00008437; 3846-05-6R2 (Other: Duke legacy protocol number)
Record Dates: First submitted 2006-06-20; First posted 2006-06-21 (Estimated); Results first posted 2013-06-04 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2012-02

CONDITIONS: Affective Disorders
Keywords: Psychotic
MeSH Terms: conditions — Mood Disorders; Mental Disorders | interventions — ziprasidone; Sertraline; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ziprasidone (Active Comparator): Subjects in this arm received ziprasidone with a placebo to maintain the blind
  Interventions: Drug: Ziprasidone
- Sertraline/Haloperidol (Active Comparator): Subjects in this arm received a combination of sertraline and haloperidol with a placebo to maintain the blind. Sertraline dosage was 150-200mg/day and haloperidol was 6-8mg/day based on tolerance.
  Interventions: Drug: Sertraline; Drug: Haloperidol

INTERVENTIONS:
Drug: Ziprasidone — Target dosage 120-160mg/day based on tolerance
  Other Names: Geodon
  Arms: Ziprasidone
Drug: Sertraline — Target dosage 150-200mg/day based on tolerance.
  Other Names: Zoloft
  Arms: Sertraline/Haloperidol
Drug: Haloperidol — Target dosage 6-8mg/day based on tolerance.
  Other Names: Haldol
  Arms: Sertraline/Haloperidol

SUMMARY:
The purpose of this study is to compare ziprasidone (Geodon) monotherapy for the treatment of psychotic major depression (PMD)with an antidepressant/antipsychotic combined therapy.

DETAILED DESCRIPTION:
Psychotic depression is a well-established DSM-IV diagnostic subtype indicating the presence of hallucinations and/or delusions as part of the clinical presentation. Currently the treatment of choice for psychotic depression is either electroconvulsive therapy or combination of antipsychotic and antidepressant medications. Ziprasidone will be compared to standard of care treatment comprising a combination of an antidepressant, sertraline and an antipsychotic, haloperidol, over a 12-week period. An additional 12-week extension phase is also included for responders to the initial study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged 18-70 years
* If female, must state willingness to use medically accepted methods of birth control (if of reproductive age) and have negative pregnancy test
* Ability to understand study procedures and provide written informed consent
* A DSM-IV diagnosis of Major Depressive Disorder, with psychotic features, based on the Structured Clinical Interview for DSM-IV (SCID)
* Hamilton Depression Rating Scale score (21-item HDRS) greater than or equal to 22

Exclusion Criteria:

* A current or lifetime DSM-IV diagnosis of Bipolar Disorder, Schizophrenia or Schizoaffective Disorder
* A DSM-IV diagnosis of alcohol or substance abuse or dependence within 3 months of study entry
* A QTc greater than 460 msec or an abnormal EKG (except minor abnormalities considered by the site investigator to be clinically insignificant)
* A heart rate less than or equal to 50
* A personal or family history of QTc
* Any current or past history of syncope
* Concurrent treatment with medications associated with prolongation of the QTc
* Concurrent treatment with medications that may affect magnesium or potassium, such as diuretics
* Any acute, unstable or serious medical illness (eg, AIDS, history of seizures, history of CVAs).
* Baseline blood chemistries that are outside local reference ranges and which are felt clinically significant by the site investigator, or a potassium, magnesium or calcium level outside of local reference ranges or liver function tests that are greater than 20% above the upper limit of local reference ranges. If magnesium and/or potassium are below the lower limit of the local laboratory norm, they may be repeated and rechecked during the screening phase, and if within laboratory norms, the subjects may be included.
* History of unstable cardiovascular disease
* A significant risk of suicide in the judgement of the site investigator
* A history of allergy or hypersensitivity to haloperidol, sertraline or ziprasidone
* Any history of neuroleptic malignant syndrome
* Treatment with sertraline or ziprasidone within 30 days of study entry
* History of recent treatment with any long acting psychotropic medications
* Treatment with a MAO-inhibitor within 14 days of study entry
* Treatment with an investigational drug within 30 days of study entry
* Current use of carbamazepine, nefazodone, ketoconazole or erythromycin
* A positive pregnancy test
* A positive drug screen unless attributable to a prescribed medication (e.g. benzodiazepines)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-04; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Cassidy, MD, Principal Investigator — Duke University; George Simpson, MD, Principal Investigator — University of Southern California; Ranga Krishnan, MD, Principal Investigator — Duke University; Sumant Khanna, MD, Principal Investigator — National Institute of Mental Health and Neuroscience; Adel Elsheshai, MD, Principal Investigator — Alexandria University
Locations (3):
- University of Southern California, Los Angeles, California, United States
- Alexandria University, Alexandria, Egypt
- National Institute of Mental Health and Neuroscience, Bangalore, India

RESULTS

PARTICIPANT FLOW:
Groups:
- Ziprasidone: Target dosage of 120-160mg/day based on tolerance.
- Sertraline/Haloperidol: Target dosage of 150-200mg/day for sertraline and 6-8mg/day for haloperidol.
Period: Overall Study
Arm/Group | Ziprasidone | Sertraline/Haloperidol
Started | 35 | 37
Completed | 27 | 28
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone | Sertraline/Haloperidol | Total
Number analyzed (Participants) | 35 | 37 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 37 | 72
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (8.7) | 35.9 (12.0) | 36.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 14 | 17 | 31
Region of Enrollment [Number; unit: participants]
  Egypt | 14 | 15 | 29
  United States | 3 | 5 | 8
  India | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: 21 Item Hamilton Depression Rating Scale
Description: The scale rates 21 symptoms related to major depression. A total score of 0-7 is considered to be normal, scores of 20 or higher indicate moderately severe depression. Total scores range from a minimum of 0(not ill) to a maximum of 64 (severely ill).
Time Frame: 12 week
Population: Number of participants was ITT and imputed by LOCF
Measure: Mean (Standard Deviation); unit: Units on Hamilton Depression Scale
Arm/Group | Ziprasidone | Sertraline/Haloperidol
Number analyzed (Participants) | 35 | 37
Units on Hamilton Depression Scale | 13.6 (8.3) | 11.0 (7.7)

2. Primary Outcome: Clinical Global Impression Improvement Scale
Description: A 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. Overall the scale goes from a minimum of 1(very much improved) to a maximum of 7(very much worse).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a Clinical Impressions Scale
Arm/Group | Ziprasidone | Sertraline/Haloperidol
Number analyzed (Participants) | 35 | 37
units on a Clinical Impressions Scale | 3.1 (2.0) | 2.5 (1.6)

3. Primary Outcome: Brief Psychiatric Rating Scale at 12 Weeks
Description: A rating scale used to measure psychiatric symptoms such as depression, anxiety, hallucinations and unusual behaviour. Each symptom is rated 1-7 and in this version a total of 24 symptoms are scored. Thus the total range of scores is from a minimum of 24 to a maximum of 168. Lower scores are considered better, so the minimum total score of 24 indicates someone with no psychiatric symptoms, while any score over 40 is considered at least moderately severe, with only the most severely ill patients scoring over 60.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a Psychiatric Rating scale
Arm/Group | Ziprasidone | Sertraline/Haloperidol
Number analyzed (Participants) | 35 | 37
units on a Psychiatric Rating scale | 28.7 (10.1) | 25.8 (6.5)

ADVERSE EVENTS:
Arm/Group | Ziprasidone | Sertraline/Haloperidol
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/37
Other Adverse Events (participants affected / at risk) | 28/35 | 33/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ziprasidone (N=35) | Sertraline/Haloperidol (N=37)
Death (General disorders) | 1 (1) | 0 (0) — Patient fell down well and died
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=35) | Sertraline/Haloperidol (N=37)
Extrapyramidal symptoms (Nervous system disorders) | 10 | 15
Akathisia (Nervous system disorders) | 13 | 8
Tremors (Nervous system disorders) | 4 | 9
Gastritis (Gastrointestinal disorders) | 8 | 2
Rigidity (Nervous system disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No